CLINICAL TRIAL: NCT02019381
Title: The Effects of Vitamin D and Calcium Supplementation at Tolerable Upper Limit Doses on Calcium Metabolism in Postmenopausal White Women.
Brief Title: Study the Effects of Vitamin D and Calcium Supplementation at Tolerable Upper Limit Doses on Calcium Metabolism.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, John F. Aloia, MD, Chief Academic Officer, MD, Endocrinology., Winthrop University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 13005
Record Dates: First submitted 2013-09-12; First posted 2013-12-24 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Delusion of Reference
MeSH Terms: interventions — Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endocrine Society UL Dosage Vitamin D (Other): Participants will be randomly assigned vitamin D + calcium dose based on Endocrine Society Upper limit guidelines. And given 10,000IU Vitamin D + 1200mg Calcium (600IU Placebo Vitamin D, in addition to two calcium tablets of 600mg) each to be taken per day.
  Interventions: Dietary Supplement: Endocrine Society UL Dosage Vitamin D; Dietary Supplement: Calcium
- Institute of Medicine Dosage Vitamin D (Other): Participants will be randomly assigned Vitamin D dose based on IOM guidelines; calcium dose will be as per IOM upper limits. And will receive 600 IU Vitamin D + 1,200 mg of calcium tablets to be taken per day.
  Interventions: Dietary Supplement: Institute of Medicine Dosage Vitamin D; Dietary Supplement: Calcium

INTERVENTIONS:
Dietary Supplement: Endocrine Society UL Dosage Vitamin D — Endocrine Upper limit arm will get 10,000IU Vitamin D and 1200mg Calcium
  Arms: Endocrine Society UL Dosage Vitamin D
Dietary Supplement: Institute of Medicine Dosage Vitamin D — IOM arm will get 600 IU Vitamin D and 1,200 mg Calcium
  Arms: Institute of Medicine Dosage Vitamin D
Dietary Supplement: Calcium — 1200mg of CaCO3 supplementation will be given to each participant in both groups

SUMMARY:
Recently two distinguished committees, Institute of Medicine (IOM) and The Endocrine Society have proposed different intake guidelines for Calcium and Vitamin D. We wish to compare the effects of both of them on calcium metabolism and bone turnover. We propose a one year randomized double blinded study for the same.

DETAILED DESCRIPTION:
The specific aims of this study proposal are to determine the following:

1. To compare the two different intake guidelines for Calcium and Vitamin D Supplementation at its recommended tolerable upper limit on serum and urinary calcium in white postmenopausal Women.
2. Compare the effects above mentioned two intake guidelines on Vitamin D metabolism [25(OH)D, 1,25(OH)2D] and bone turnover.

Participants will be randomly assigned to Group A or Group B based on different dosages of study medications.

Group A: 10,000 IU (International Units)Vitamin D + Placebo (sugar pill) 600IU Vitamin D + Two pills Calcium containing 600mg calcium each.

Group B: 600 IU Vitamin D + Placebo (sugar pill) 10,000 IU Vitamin D

+ Two pills Calcium containing 600mg calcium each.

In addition to the calcium supplements, they will guide to include approximately 800mg of calcium in their daily diet.

At visit 2, fasting blood and spot urine will be collected. A urinal will be dispensed for collection of 24-hour urine for urinary calcium to be brought in next day. Study medication will be dispensed and participants will be asked not to discard unused medications and to bring all study medications next study visit.

Visit 3, 4, 5, 6 will essentially be the same as visit 2, with subjects returning unused study medication and given new tablets each visit. Except on visit 6 no further study medications will be dispensed, after collecting the previous supply.

Food frequency questionnaires will be filled out at the initial visit and final visit. Diet will be assessed using 3-day diet history form and Nutrition Pro analysis software. Patients will be asked to refrain from taking other Vitamin D supplements and to continue their usual calcium intake.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy White women aged 50 and older who have been postmenopausal for at least 2 year (i.e. absence of menstrual period for a period of 24 months or more).
2. Willingness to discontinue self-administration of vitamin D and calcium supplements. Participants must be at least three months off supplements before starting the study.
3. Willingness to take study medications and participate in study for one year.
4. Written informed Consent Signed.
5. Patients with hypertension and diabetes stable for last three months.

Exclusion Criteria:

1. History of hypercalciuria (24-hour urinary calcium excretion >250 mg), hypercalcemia (serum calcium >10.6), nephrolithiasis and active sarcoidosis will be excluded.
2. Serum 25-hydroxyvitamin D level >80 nmol/L or history of primary hyperparathyroidism.
3. Dietary calcium intake of >2000mg/day will be excluded
4. Use of medication that influences bone or vitamin D metabolism (e.g. anticonvulsant medications, glucocorticoids, Highly Active AntiRetroviral Therapy [AIDS treatment], antirejection medications, chronic use of steroids, high dose diuretics)
5. Treatment with Hormone replacement therapy, Selective Estrogen Receptor Modulators, Calcitonin, Parathyroid hormone , androgens, bisphosphonates, phosphate or anabolic steroids 6 months prior to the study.
6. Use of systemic steroids (oral or intravenous) within the last year at an average dose of more than 5mg/day of oral prednisone or an equivalent for a period of three months or more prior to screening.
7. Chronic medical illness including Chronic liver disease, uncontrolled diabetes mellitus; recent history of myocardial infarction or heart failure; newly diagnosed or active malignancy; uncontrolled hypertension; obesity (BMI>35 kg/m2); malabsorption, anemia, leukemia, or other hematologic abnormalities; lupus, rheumatoid arthritis, sarcoidosis, or other rheumatologic disease; chronic kidney disease, metabolic bone disease.
8. Unexplained weight loss of >15% during the previous year or history of anorexia nervosa
9. > 1 pack per day tobacco use or > 2 alcoholic beverages per day
10. Unwillingness to forego self-administration of vitamin D and calcium-containing supplements.
11. Participation in another investigational trial in the past 30 days prior to the screening evaluation
12. Significant deviation from normal in medical history, physical examination, or laboratory tests as evaluated by the primary investigator.
13. Patients with unstable hypertension or diabetes.

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Compare the effects of 10000 IU/day vitamin D plus 2,000 mg/day calcium versus 600 IU/day vitamin D plus 2,000 mg/day calcium on incidence of hypercalciuria (spot urine calcium:creatinine ratio, 24-hour urine calcium). | One year
  Endocrine society has recommended tolerable upper limit or a dose with no adverse events as 10,000IU of Vitamin D and 2000 mg/day of calcium. Our study will test the safety/ efficacy of this recommendation.

SECONDARY OUTCOMES:
Compare the effects of 10,000 IU/day vitamin D plus 2,000 mg/day calcium versus 600 IU/day vitamin D plus 2,000 mg/day calcium on vitamin D metabolism [25(OH)D, 1,25(OH)2D], and bone turnover. | One year
  To test safety/efficacy of The Endocrine Society recommendations on Bone turnover.

CONTACTS AND LOCATIONS:
Overall Officials: John Aloia, MD, Principal Investigator — Winthrop UH; Mageda Mikhail, MD, Study Director — Winthrop UH
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aloia JF, Katumuluwa S, Stolberg A, Usera G, Mikhail M, Hoofnagle AN, Islam S. Safety of calcium and vitamin D supplements, a randomized controlled trial. Clin Endocrinol (Oxf). 2018 Dec;89(6):742-749. doi: 10.1111/cen.13848. Epub 2018 Oct 1. PMID 30180273